CLINICAL TRIAL: NCT02371265
Title: Early ART Initiation Among HIV-positive Pregnant Women in Central Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Health Alliance International (Other); Beira Operations Research Center, Mozambique Ministry of Health (Unknown)
Responsible Party: Principal Investigator, James Pfeiffer, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 42773; 1R01HD074557-01 (NIH)
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: HIV
Keywords: HIV; Mozambique; antenatal care; adherence; retention; pregnancy; HIV-positive mothers retained in ART after 90 days

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adherence and retention intervention (Experimental): Implementation of adherence and retention package
  Interventions: Other: Adherence and retention package
- Control (No Intervention): Clusters continue without intervention package

INTERVENTIONS:
Other: Adherence and retention package — Based on formative research findings, the following core components of the B+ study intervention have been designed and will be stepped in at the study sites to improve early retention in care and adherence:
  * Workflow modification: 1) Redefinition of key roles of MCH nurses and task shifting to community health workers (CHW's), and 2) enhanced patient tracking via improved management of registries/charts;
  * Adherence and retention package: 1) Creation of "Adherence Committees" at each site to coordinate and systematize patient follow-up, 2) active patient follow-up and home visits by community health workers (CHWs or activistas), 3) use of text messaging to patients by MCH nurses, 4) improved and intensified counseling coordinated with active CHW and text follow-up, and 5) intensified and improved Option B+ training and supportive supervision.
  Arms: Adherence and retention intervention

SUMMARY:
The overall objective of the study is to develop and test a pilot intervention in central Mozambique to implement the new WHO "Option B+" guidelines that seek to increase the proportion of HIV-positive pregnant women in six antenatal care clinics who start antiretroviral therapy (ART) prior to delivery, and are retained in care after 90- days.

DETAILED DESCRIPTION:
For over 10 years, services to prevent maternal to child HIV-1 transmission (PMTCT) have been scaled-up and integrated into antenatal care (ANC) in the national health system across Mozambique. In 2004, scale-up of anti-retroviral treatment (ART) also began in Mozambique and is now provided at hundreds of health units. In 2010, the World Health Organization developed new treatment guidelines, termed "Option B" that emphasized early initiation of ART in antenatal care for all HIV-positive pregnant women. In 2012, the WHO issued a programmatic update endorsing a third option termed "Option B+" in which HIV positive pregnant women initiate ART during pregnancy regardless of disease progression and continue treatment for life.

The new "Option B+" approach has been adopted by the Ministry of Health (MoH) in Mozambique and is in the early phases of implementation. As in many African settings, numerous health system factors present major challenges to successful adoption of the guidelines. In Mozambique, ANC and HIV testing coverage is high but there is substantial loss-to-follow-up (LTFU) at successive stages in the treatment cascade, limited counseling for women and many barriers to actively tracking those women lost to follow-up. Early Ministry of Health data suggests significant challenges remain for long-term adherence for women started on ART via the new Option B+ framework in Manica and Sofala provinces and throughout Mozambique.

The successful implementation of new WHO guidelines therefore requires major streamlining of links among ANC, PMTCT, and ART services. The overall objective of this study is to develop and test a pilot intervention in central Mozambique to implement the new WHO guidelines, and increase the proportion of HIV-positive pregnant women in target ANC clinics who start ART prior to delivery, without reducing ART adherence in the first 3 months of therapy. The intervention will emphasize a WHO defined "Option B+" approach; HIV-positive mothers will be referred for ART at the time they receive a positive HIV test result in their first ANC visit. The project utilizes an innovative formative research process, which has already been completed, and a stepped wedge implementation science design to evaluate the intervention. The entire study is being conducted in close collaboration with the Center for Operations Research in Beira (known by its Portuguese acronym as CIOB) that is one of three research centers in Mozambique managed by the MOH National Institute of Health (the research arm of the MoH).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who test HIV-positive in antenatal care services at target health facilities

Exclusion Criteria:

* Pregnant women who arrived at health facilities who already have tested positive
* HIV-positive pregnant women who cannot start ART

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 761 (Actual)
Dates: Start 2012-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Retention at 30 days | 45 days
  The primary outcome measure for Aim 3 is the proportion of HIV-positive pregnant women tested at the participating ANC sites that successfully initiates appropriate ART and returns for their scheduled 30-day visit for pharmacy refill and evaluation within 45 days.
Adherence at 90 days | 90 days
  The primary outcome measure for Aim 4 is the ART adherence rate through 90 days after ART initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Chapman, PhD, Principal Investigator — University of Washington
Locations (1):
- Beira Operations Research Center, Beira, Sofala, Mozambique

REFERENCES:
- [Derived] Cowan JF, Micek M, Cowan JF, Napua M, Hoek R, Gimbel S, Gloyd S, Sherr K, Pfeiffer JT, Chapman RR. Early ART initiation among HIV-positive pregnant women in central Mozambique: a stepped wedge randomized controlled trial of an optimized Option B+ approach. Implement Sci. 2015 Apr 30;10:61. doi: 10.1186/s13012-015-0249-6. PMID 25924668